CLINICAL TRIAL: NCT02936375
Title: The Effect of Iguratimod on Active Lupus Nephritis, the IGeLU Study: a Randomized Controlled Trial
Brief Title: The Iguratimod Effect on Lupus Nephritis (IGeLU)
Acronym: IGeLU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2016]128k
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Lupus Nephritis
Keywords: lupus; nephritis; iguratimod
MeSH Terms: conditions — Lupus Nephritis; Nephritis | interventions — iguratimod; T 614; Clinical Coding; Cyclophosphamide; Azathioprine; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iguratimod (Experimental): Patients will receive iguratimod over the whole follow-up, combined with steroids, as well as auxiliary treatment (such as vitamin D, gastrointestinal agents, blood pressure medications, if any)
  Interventions: Drug: Iguratimod; Drug: Steroids
- Cyc+AZA (Active Comparator): Patients will receive cyclophosphamide in the first half of study (usually to 24 weeks), followed with azathioprine till the end of follow-up. Patients will also receive steroids as combinational therapy, as well as auxiliary treatment (such as vitamin D, gastrointestinal agents, blood pressure medications, if any)
  Interventions: Drug: Cyclophosphamide; Drug: Azathioprine; Drug: Steroids

INTERVENTIONS:
Drug: Iguratimod — 25mg twice a day, orally administrated
  Other Names: T-614 (code name); Iremod (brand name)
  Arms: Iguratimod
Drug: Cyclophosphamide — 1g/m², every 4 weeks, intravenous
  Arms: Cyc+AZA
Drug: Azathioprine — 2mg/kg·d, once a day, orally administrated
  Arms: Cyc+AZA
Drug: Steroids — Prednisone, methylprednisolone or prednisonlone, once a day, orally administrated. Steroids should be 1mg/kg·d in the beginning four weeks, then tapered 5-10mg/d every two weeks till 30mg/d, then tapered 2.5-5mg/d every two weeks. After 24 weeks of follow-up, a patient should receive steroids no more than 10mg/d. Patients may receive temporal high dose of steroids (1mg/kg·d) because of symptoms outside of kidney, for no more than two weeks. All the dosage of steroids above is calculated by prednisone.

SUMMARY:
This study is a 52-week, randomized, open, active-controlled trial of patients with active diffused lupus nephritis, to assess the efficacy and safety of a novel chemical synthetic agent iguratimod. The subjects will randomly receive iguratimod or cyclophosphamide followed with azathioprine, both combined with steroids.

ELIGIBILITY:
Inclusion Criteria:

* Active lupus nephritis:

  * Fulfill ACR classification criteria (2009) for SLE
  * Proteinuria ≥1g/24h at screening
  * Nephritis of class III, IV, V, III+IV or IV+V, confirmed by renal pathology within 90 days prior to screening
* Body weight ≥40kg
* SLE-2K score ≥8
* Agreement of contraception
* Informed consent obtained

Exclusion Criteria:

* Active severe SLE-driven renal disease or unstable renal disease at screening
* Active severe or unstable neuropsychiatric SLE
* Clinically significant active infection including ongoing and chronic infections
* History of receiving cyclophosphamide, azathioprine, tacrolimus , mycophenolate moetil or rituximab treatment with 90 days prior to screening
* History of human immunodeficiency virus (HIV)
* Confirmed Positive tests for hepatitis B or positive test for hepatitis C
* Active tuberculosis
* Live or attenuated vaccine within 4 weeks prior to screening
* Subjects with significant hematologic abnormalities
* Abnormal liver function test at screening (ALT, AST or total bilirubin over 2 fold of upper normal level
* History of peptic ulcer or GI bleeding; treatment with warfarin or other anticoagulants within last 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
renal remission rate | Week 52

SECONDARY OUTCOMES:
Renal remission rate | Week 24
Renal flare rate | Week 52
Number of participants with treatment-related adverse events | Week 52
  adverse events are assessed by CTCAE v4.0
SLEDAI-2K score | Week 52
  SLE SLE disease activity index (2000)
BILAG score | Week 52
  British Isles lupus assessment group score
PGA | Week
  Patient general assessment

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, MD, Principal Investigator — RenJi Hospital
Locations (2):
- China (2):
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Yan Q, Du F, Kang Y, Ye P, Wang X, Xu J, Tang J, Wang N, Jiang G, Li Z, Wang X, Xue Q, Huang X, Zhang X, Zhou Y, Dai M, Bao C. Comparison of iguratimod and conventional cyclophosphamide with sequential azathioprine as treatment of active lupus nephritis: study protocol for a multi-center, randomized, controlled clinical trial (iGeLU study). Trials. 2021 Aug 11;22(1):530. doi: 10.1186/s13063-021-05475-3. PMID 34380536